CLINICAL TRIAL: NCT02143752
Title: Meriter Mindfulness Training for Smokers Program and Study
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-001; 2012-001 (Other Grant/Funding Number: Meriter Hospital)
Record Dates: First submitted 2013-01-17; First posted 2014-05-21 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2015-04

CONDITIONS: Smoking
Keywords: Smoking; Tobacco; Addiction; Mindfulness; Meditation
MeSH Terms: conditions — Smoking; Behavior, Addictive | interventions — Mindfulness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mindfulness: Smokers enter a Mindfulness Training for Smokers course
  Interventions: Behavioral: Mindfulness
- Quit Line: Smokers attempt smoking cessation with the help of the Wisconsin Tobacco Quit Line
  Interventions: Behavioral: Quit Line

INTERVENTIONS:
Behavioral: Mindfulness — Group behavioral intervention using mindfulness to help smokers quit smoking
  Other Names: Mindfulness Training for Smokers
  Groups: Mindfulness
Behavioral: Quit Line — see arm
  Other Names: see arm
  Groups: Quit Line

SUMMARY:
The Meriter Smoking Cessation Study tests participants in the Meriter Smoking Cessation Program. Meriter Hospital and clinic patients will be recruited into the Meriter Smoking Cessation Program. The Meriter Smoking Cessation Program has two interventions, the Mindfulness Training for Smokers (MTS) intervention and the Quit Line (QL) Intervention. Study activities include one 10-minute study visit and two 5-minute survey phone calls.

DETAILED DESCRIPTION:
The Meriter Smoking Cessation Study tests participants in the Meriter Smoking Cessation Program. Meriter Hospital and clinic patients will be recruited into the Meriter Smoking Cessation Program. The Meriter Smoking Cessation Program has two interventions, the Mindfulness Training for Smokers (MTS) intervention and the Quit Line (QL) Intervention. Study activities include one 10-minute study visit and two 5-minute survey phone calls.

MTS: Mindfulness Training for Smokers Intervention. This is the 7-week quit smoking intervention developed by the PI.

QL: Quit Line Intervention. This is a program starting at makes use of the Wisconsin Tobacco Quit Line.

Meriter Smoking Cessation Program: A program offering the MTS and QL interventions to smokers at Meriter Hospital and Clinics.

Meriter Smoking Cessation Study: This is a study comprised of 2 phone surveys and 1 study visit that tests participants in the MTS and QL intervention. Participants in the Meriter Smoking cessation program will have the opportunity to decide if they would like to be in the study.

ELIGIBILITY:
Inclusion Criteria:

* everyday smoker

Exclusion Criteria:

* current alcohol or other drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be drawn from the Meriter Smoking Cessation Program, which is made up of two interventions: the Mindfulness Training for Smokers (MTS) intervention and the Quit Line (QL) Intervention
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
biochemically confirmed post treatment smoking abstinence | 10 days post quit
  Carbon monoxide levels are obtained 10 days post quit. CO under 7 = abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: James M Davis, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Meriter Hospital and Medical Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Davis JM, Mills DM, Stankevitz KA, Manley AR, Majeskie MR, Smith SS. Pilot randomized trial on mindfulness training for smokers in young adult binge drinkers. BMC Complement Altern Med. 2013 Sep 3;13:215. doi: 10.1186/1472-6882-13-215. PMID 24006963
- See also: Pilot randomized trial on mindfulness training for smokers in young adult binge drinkers — http://www.ncbi.nlm.nih.gov/pubmed/24006963